CLINICAL TRIAL: NCT04755842
Title: Tricuspid Regurgitation Hamburg Cohort
Acronym: TRUTH
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: TRUTH
Record Dates: First submitted 2021-02-07; First posted 2021-02-16 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Standardized methods for sample collection, processing, and storage, as well as appropriate storage facilities, are established and managed in accordance with the highest scientific and ethical standards. To ensure uniformity, quality, and reproducibility for the collection, processing, and storage of biomaterial, standard operating procedures (SOPs) are implemented.
  The following biomaterial will be sampled for additional biobanking within study visits, as described above:
  * Blood (whole blood, serum, plasma (EDTA, citrated,), DNA, RNA, washed erythrocytes
  * Urine
  * Tissue/ cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tricuspid regurgitation (TR) is frequent and has been directly related to high mortality rates. The pathophysiology of TR is mainly functional as it occurs predominantly in the context of left-sided heart disease, pulmonary hypertension, or atrial fibrillation. Surgery is currently the primary treatment option in patients with functional TR. However, isolated tricuspid valve surgery is associated with an intolerable high risk of operative mortality and poor outcomes. New transcatheter options could be used in high-surgical risk patients. However, with often severely dilated annuli with a non-planar and elliptical shape, absence of calcification, and proximity of structures, the tricuspid valve anatomy poses many challenges.

Predictors of outcome are yet to be defined in patients with TR in order to improve risk prediction for the different treatment modalities (medical, surgical, interventional). The Tricuspid Regurgitation Hamburg Cohort (TRUTH) aims to monitor patients with relevant TR, irrespective of the underlying etiology or therapeutic approach. In addition to available evidence from previously published clinical trials, elaborate prospective clinical registries, such as TRUTH, that monitor clinical routine and current practice, will be of significant importance to further enhance therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent in accordance with Good Epidemiological Practice and local legislation.
* Individuals over the age of 18 years.
* Patients with clinically relevant tricuspid regurgitation (≥ severe TR, at least Grade III of V)

Exclusion Criteria:

* Insufficient knowledge of the German language, to understand study documents and interview without translation
* Physical or psychological incapability to cooperate in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Tricuspid Regurgitation Hamburg Cohort (TRUTH) aims to monitor patients with severe TR, irrespective of the underlying etiology or therapeutic approach.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 6-60 months
  Incidence of death from any cause.
Cardiovascular mortality | 6-60 months
  Incidence of cardiovascular death, defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Rehospitalization for congestive heart failure | 6-60 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization, e.g. as assessed by patient interviews.
Unplanned tricuspid valve intervention | 6-60 months
  Incidence of unplanned surgical or transcatheter re-intervention, heart transplantation or assist device implantation, e.g. as assessed by patient interviews.
Tricuspid regurgitation severity | 6-60 months
  Tricuspid regurgitation (TR) severity measured by transthoracic and transesophageal echocardiography. Assessment of TR severity according to current recommendations for valvular heart disease.

SECONDARY OUTCOMES:
Change in 6-minute-walking-test (6MWT) distance | 6-60 months
  6MWT will be performed by all participants at baseline and at follow-up visits.
Change in quality of life | 6-60 months
  Quality of life will be assessed by a standardized questionnaire [Kansas City Cardiomyopathy Questionnaire [KCCQ]) in all participants at baseline and at follow-up visits (or by phone interviews).
  The score is represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and a score of 100 indicates no symptoms, no limitations, and excellent quality of life.
Change in New York Heart Association (NYHA) functional class | 6-60 months
  New York Heart Association [NYHA] functional class (I-IV) will be assessed in all participants at baseline and at follow-up visits (or by phone interviews).
  NYHA Class I: No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  NYHA Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  NYHA Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  NYHA Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kalbacher, MD, Principal Investigator — University Heart and Vascular Center Hamburg; Edith Lubos, MD, Principal Investigator — University Heart and Vascular Center Hamburg
Locations (1):
- University Heart and Vascular Center Hamburg, Hamburg, Germany